CLINICAL TRIAL: NCT05982444
Title: Long Term Post-operative Effectiveness and Morbidity of Rezum Therapy for Benign Prostatic Hyperplasia
Brief Title: Long Term Follow up of Water Vapor Thermal Therapy (Rezum) for Benign Prostatic Hyperplasia (BPH)
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Helwan University (Other)
Responsible Party: Principal Investigator, Mahmoud Mohammed Elsaid Ali Elshahawy, Principal Investigator, Faculty of medicine, Helwan University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 30-2023
Record Dates: First submitted 2023-07-24; First posted 2023-08-08 (Actual); Last update posted 2025-06-27 (Actual); Status verified 2025-06

CONDITIONS: Benign Prostatic Hyperplasia; Lower Urinary Track Symptoms
Keywords: water vapor thermal therapy
MeSH Terms: conditions — Prostatic Hyperplasia

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- patient treated by rezum procedure (Other): patients had benign prostatic hyperplasia and treated by rezum procedure from 2 to 4 years included in the study
  Interventions: Procedure: water vapor thermal therapy (Rezum) for prostate

INTERVENTIONS:
Procedure: water vapor thermal therapy (Rezum) for prostate — all patients underwent rezum therapy for bph are evaluated for its effectiveness for long period
  Other Names: Prostate steam treatment (Rezum) for benign prostatic hyperplasia (BPH)

SUMMARY:
This study aims to assess the effectiveness and morbidity of water vapor thermal therapy (Rezūm therapy) for benign prostatic hyperplasia (BPH). Data will be collected and analyzed from patients treated by Rezūm and followed up for 4 years prior to evaluating clinical outcomes.

DETAILED DESCRIPTION:
The investigators will conduct a retrospective study evaluating patients treated with water vapor thermal therapy (Rezūm therapy) for BPH and followed up for4 years. The primary objectives are to assess the long-term effectiveness and morbidity rates associated with the procedure. Data collected will include urinary symptom scores, sexual function, and any treatment-related complications.

ELIGIBILITY:
Inclusion Criteria:

* patients underwent rezum procedure for benign prostatic hyperplasia from 2 to 4 years

Exclusion Criteria:

* previous prostatic intervention
* concurrent urological morbidity like urethral stricture
* neurological disease like parkinson's disease

Ages: 40 Years to 80 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — the disease is conclusive for men
Enrollment: 86 (Actual)
Dates: Start 2021-03-01 (Actual); Primary Completion 2025-03-01 (Actual); Study Completion 2025-05-01 (Actual)

PRIMARY OUTCOMES:
change in prostate volume | 4 years
  Prostate volume will be measured via transrectal ultrasound.
hange in International Prostate Symptom Score (IPSS) | 4 years
  IPSS is a questionnaire evaluating urinary symptoms. Scores ranging from 0 to 7 indicate mild symptoms, from 8 to 19 moderate symptoms, and from 20 to 35 severe symptoms.
international index of erectile function (IIEF) | 4 years
  IIEF is a questionnaire evaluating sexual function. Scores ranging from 5 to 7 indicate severe symptoms, 8 to 11 moderate symptoms, 12 to 16 mild to moderate symptoms, 17 to 21 mild symptoms, and 22 to 25 no erectile dysfunction
Change in Post-Void Residual Urine | 4 years
  Residual urine volume measured after urination using pelvic ultrasound.

SECONDARY OUTCOMES:
Retreatment Rate Following Rezūm Therapy | 4 years
  Number of participants requiring additional treatment for BPH after Rezūm therapy.
complication rate | 4 years
  incidence of complications post procedure during follow-up

CONTACTS AND LOCATIONS:
Locations (1):
- Faculty of Medicine Helwan University, Helwan, Cairo Governorate, Egypt

IPD SHARING:
Plan to Share IPD: No
Patients are not permitted to post any of their personal information